CLINICAL TRIAL: NCT02659449
Title: Assessing the Impact of Different Compression of the Hand (Made to Measure Gloves / Compression Bandaging) Versus Free Hand on the Implementation of the Precision Grip
Brief Title: Assessing the Impact of Different Compression of the Hand Versus Free Hand on the Implementation of the Precision Grip
Acronym: EvICoMaB
Status: Terminated | Type: Observational
Why Stopped: No inclusion
Sponsor: Hôpital Léon Bérard (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00381-41.V1.2
Record Dates: First submitted 2015-10-27; First posted 2016-01-20 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Burned Hands
Keywords: hands
MeSH Terms: interventions — Compression Bandages

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: made to measure compression gloves — Patients achieve tests with compression glove
  Other Names: gloves of medical Z laboratory
Device: Compression bandaging — Patients achieve tests with compression bandaging
  Other Names: Coheban
Other: Free Hands — Patients achieve tests without device

SUMMARY:
The purpose of this study is to determine the impact of compressing therapy on the dexterity of burned hands using evaluating hand function tests (Box and block / Purdue Peg Board / Jamar's test)

DETAILED DESCRIPTION:
Patients with burned hands will realise prehension test to explore dexterity of hand when they wear compressive's treatments and with free hands.

Each patient will realise each test with all conditions (free hands/ made to measure gloves/ compressive bandaging).

Running order of test and condition is randomly defined. Each patient realized this tests under the care and devices used at usual care. Realisation of this tests are not influenced by the study. Patient realised this tests during reeducation.

ELIGIBILITY:
Inclusion Criteria :

* Patient admitted from Leon Bérard Hospital
* Burn hand with 2nd or 3nd degree depp
* Dominant hand if bilateral's burning
* Patients requiring compression of the hand
* Patient receiving final compression gloves since seven days ± two days weekend
* Patient affiliated to a social security

Exclusion Criteria :

* No burning of the hand
* contraindication for the use of compression
* Incompatible articular balance with achievement tests
* Patients already included in a second study
* Minor patient or pregnant woman
* Presence of cognitive disorder, preventing the achievement of tests
* Guardianship or individual under the protection of a conservator
* Patients not receiving social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with burned hands
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2016-07-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Box and Block test | mesure will be realised three time : 48h - 96h -144 hours after inclusion
  A rectangular box that is divided into two square compartments of equal dimension by means of a partition. One hundred and fifty, wooden cubes are placed in one compartment or the other. The individual move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds.
  The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period.
  The measure will be implemented for each compressive medical device and free hand (three time for each patient). Interval of 24h between each compressive.
  Measure will be realised at end of test when hand's cicatrisation will be obtained and after a time lag of 7 days after receipt of definitive compressive gloves.
  The measure will be realised every two days during one week (duration of study after inclusion of patient) after hand's evaluation by the investigator.
Purdue Pegboard test | mesure will be realised three time: 48h - 96h -144 hours after inclusion
  The Purdue Pegboard Test is a rectangular board with 2 sets of 25 holes running vertically and 4 concave cups at the top. Small metal pegs are placed in the cup on the side being tested, with subjects asked to remove the pegs and place them vertically in the holes as rapidly as possible. The number of pegs placed in 30 seconds is scored.
  The measure will be implemented for each compressive medical device and free hand (three time for each patient). Interval of 24h between each compressive.
  Measure will be realised at end of test when hand's cicatrisation will be obtained and after a time lag of 7 days after receipt of definitive compressive gloves.
  the measure will be realised every two days during one week (duration of study) after hand's evaluation by the investigator
Jamar's Test | mesure will be realised three time :48h - 96h -144 hours after inclusion
  A Hand Dynamometer is used for testing hand grip strength. The measure will be implemented for each compressive medical device and free hand (three time for each patient). Interval of 24h between each compressive.
  Measure will be realised at the hand of the test when hand's cicatrisation will be obtained and after a time lag of 7 days after receipt of definitive compressive gloves.
  the measure will be realised every two days during one week (duration of study) after hand's evaluation by the investigator

SECONDARY OUTCOMES:
Quick DASH test | 24 hours after inclusion
  This questionnaire asks about your symptoms as well as your ability to perform certain activities.
  Quick DASH test is realised 1st day after inclusion of patient on EvICoMaB clinical study and one day before realisation of hand's tests (second day of study) . The measure is obtained at end of questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Chavineau-Mortelette, MedD, Principal Investigator — Léon Bérard Hospital
Locations (1):
- Leon Berard hospital, Hyères, PACA, France